CLINICAL TRIAL: NCT03969277
Title: The Effectiveness of Graded Motor Imagery Training in Elbow Limitation
Brief Title: Graded Motor Imagery in Elbow Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 141001
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2021-06

CONDITIONS: Elbow Fracture; Limitation, Mobility; Pain, Postoperative; Upper Extremity Problem
Keywords: Imagery; Mirror Neurons; Immobilization; Exercise; Rehabilitation
MeSH Terms: conditions — Elbow Fractures; Mobility Limitation; Pain, Postoperative; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Graded Motor Imagery (Experimental): Each subject in the Graded Motor Imagery group will receive a treatment protocol consisting of Graded Motor Imagery, cold therapy, and home exercises.
  Interventions: Other: Graded Motor Imagery; Other: Home Exercise Program; Other: Cold Application
- Standard Rehabilitation (Active Comparator): Each subject in the Standard Rehabilitation group will receive a treatment protocol consisting of stretching and strengthening exercises, cold therapy, and home exercises.
  Interventions: Other: Standard Rehabilitation; Other: Home Exercise Program; Other: Cold Application

INTERVENTIONS:
Other: Graded Motor Imagery — The first stage of GMI includes laterality reconstruction. Patients will view and determine if the various images of body parts to image portrays the right or left side. The second stage targets activation of the primary motor cortex by imagine moving the involved body part. The final stage involves that the patient watches the unaffected body part moving in a mirror to "trick" the brain into thinking the affected body part is actually moving in a pain-free way. This will be applied for 6 weeks.
  Arms: Graded Motor Imagery
Other: Standard Rehabilitation — Shoulder, elbow and wrist AROM exercises. Elbow flexion and extension, and wrist flexion and extension stretching exercises. Elbow and wrist strengthening exercises. Grip strengthening exercises. This will be applied for 6 weeks.
  Arms: Standard Rehabilitation
Other: Home Exercise Program — Proprioception exercises for the elbow. Scapulothoracic strengthening exercises. This will be applied for 6 weeks.
Other: Cold Application — Cold application around the elbow joint for 15 minutes in every session.

SUMMARY:
This randomized-controlled trial aims to investigate the efficacy of Graded Motor Imagery (GMI) on function, pain, and range of motion (ROM) in patients with a posttraumatic stiff elbow.

DETAILED DESCRIPTION:
To investigate the efficacy of GMI on function, pain, and ROM in elbow limitation, voluntary patients with elbow limitation, aged between 20-55 years will be randomly divided into two groups: GMI group and standard rehabilitation (SR) group. Interventions will be applied for 12 sessions. The patients will be assessed before, after six-week treatment and six-week follow-up. The pain on activity, at rest and at night will be assessed with Visual Analog Scale (VAS). Pain pressure threshold of the elbow and soft tissue around the elbow will be evaluated by digital pressure algometry. ROM will be assessed with a digital goniometer. Isometric muscle strength will be measured with a handheld dynamometer of elbow flexors and extensors. Grip strength will also be assessed. Recognise™ will be used for assessing the right-left discrimination. The functional status and kinesiophobia will be evaluated by Disabilities Arm, Shoulder and Hand (DASH) and Tampa Scale for Kinesiophobia, respectively. The Global Rating of Change will be used to evaluate patient satisfaction. The Vividness of Movement Imagery Questionnaire 2 (VMIQ-2) will be used for evaluating the individuals' ability to mental imaginary.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included with

* Aged between 20 and 55 years
* Elbow fracture in the six months before the study
* Elbow limitation in flexion or extension
* Being a volunteer to participate
* Fractures should be managed with surgically
* The "Standardized Mini Mental Test" result must be at least 24 points

Exclusion Criteria:

* Malunion or Nonunion Fracture
* The occurrence of complex regional pain syndrome, peripheric nerve injury, heterotopic ossification, myositis ossification or post-traumatic ankylosing
* Non-healing wound or infection
* Previously received physiotherapy for elbow limitation
* Having any cardiovascular diseases, neurological disorders, rheumatic diseases or psychiatric diseases
* Could not adjust to the treatment
* Shoulder, elbow or wrist movement limitation in contralateral upper extremity or absence of limbs in the contralateral upper extremity
* Having severe visual loss

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Functional Status | After the six-week intervention
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH). It comprises 30 core questions and optional additional 8 questions that are scored on a 5-point Likert-type scale (no difficulty-unable). The cumulative DASH score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.

SECONDARY OUTCOMES:
Pain Intensity | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Pain Intensity | After the six-week intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Pain Intensity | 6-week follow-up
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion (AROM) Assessment | Baseline
  The elbow's and forearm's AROM, including flexion, extension, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the average value recorded.
Active Range of Motion (AROM) Assessment | After the six-week intervention
  The elbow's and forearm's AROM, including flexion, extension, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the average value recorded.
Active Range of Motion (AROM) Assessment | 6-week follow-up
  The elbow's and forearm's AROM, including flexion, extension, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the average value recorded.
Functional Status | Baseline
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH). It comprises 30 core questions and optional additional 8 questions that are scored on a 5-point Likert-type scale (no difficulty-unable). The cumulative DASH score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.
Functional Status | 6-week follow-up
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH). It comprises 30 core questions and optional additional 8 questions that are scored on a 5-point Likert-type scale (no difficulty-unable). The cumulative DASH score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.
Fear of movement (kinesiophobia) | Baseline
  Kinesiophobia of the patients will be assessed by Tampa Scale for Kinesiophobia. It is a 17-item questionnaire scored on a 4-point Likert-type scale (strongly disagree-strongly agree). The total score of the scale ranged from 17 to 68, with higher scores indicating more kinesiophobia.
Fear of movement (kinesiophobia) | After the six-week intervention
  Kinesiophobia of the patients will be assessed by Tampa Scale for Kinesiophobia. It is a 17-item questionnaire scored on a 4-point Likert-type scale (strongly disagree-strongly agree). The total score of the scale ranged from 17 to 68, with higher scores indicating more kinesiophobia.
Fear of movement (kinesiophobia) | 6-week follow-up
  Kinesiophobia of the patients will be assessed by Tampa Scale for Kinesiophobia. It is a 17-item questionnaire scored on a 4-point Likert-type scale (strongly disagree-strongly agree). The total score of the scale ranged from 17 to 68, with higher scores indicating more kinesiophobia.
Patient Satisfaction | After the six-week intervention
  Patient satisfaction regarding improvement in elbow function will be assessed by the Global Rating of Change scale. The participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly in this study.
Right-Left Discrimination | Baseline
  Right-Left Discrimination will be assessed with Recognise™ application. It tests the patients' ability to quickly and accurately recognise an image of a body area as either left or right ('Left/Right Discrimination'). The test will be repeated three times and average values will be recorded.
Right-Left Discrimination | After the six-week intervention
  Right-Left Discrimination will be assessed with Recognise™ application. It tests the patients' ability to quickly and accurately recognise an image of a body area as either left or right ('Left/Right Discrimination'). The test will be repeated three times and average values will be recorded.
Right-Left Discrimination | 6-week follow-up
  Right-Left Discrimination will be assessed with Recognise™ application. It tests the patients' ability to quickly and accurately recognise an image of a body area as either left or right ('Left/Right Discrimination'). The test will be repeated three times and average values will be recorded.
Vividness of Movement imagery Questionnaire-2 (VMIQ-2) | Baseline
  The Vividness of Movement Imagery Questionnaire-2 (VMIQ-2) will be used to measure the vividness of imagery. It comprises three subscales and 12 core questions that are scored on a 5-point Likert-type scale (Perfectly clear and as vivid (as normal vision or feel of movement) - No image at all, you only "know" that you are thinking of the skill). The subscales scores (External Visual Imagery, Internal Visual Imagery, and Kinaesthetic imagery) are ranged from 1 to 60, where the higher scores indicate a decreased ability of vividness of imagery.
Pain pressure threshold | Baseline
  Pain pressure threshold of the elbow and soft tissue around the elbow will be evaluated by digital pressure algometry. The process will be repeated three times in each direction, with the average value recorded.
Pain pressure threshold | After the six-week intervention
  Pain pressure threshold of the elbow and soft tissue around the elbow will be evaluated by digital pressure algometry. The process will be repeated three times in each direction, with the average value recorded.
Pain pressure threshold | 6-week follow-up
  Pain pressure threshold of the elbow and soft tissue around the elbow will be evaluated by digital pressure algometry. The process will be repeated three times in each direction, with the average value recorded.
Muscle strength | After the six-week intervention
  Isometric muscle strength will be measured with a handheld dynamometer for elbow flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Muscle strength | 6-week follow-up
  Isometric muscle strength will be measured with a handheld dynamometer for elbow flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Grip strength | After the six-week intervention
  Grip strength will be assessed with JAMAR hydraulic hand dynamometer. The process will be repeated three times in each direction, with the average value recorded.
Grip strength | 6-week follow-up
  Grip strength will be assessed with JAMAR hydraulic hand dynamometer. The process will be repeated three times in each direction, with the average value recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

REFERENCES:
- [Background] Mendez-Rebolledo G, Gatica-Rojas V, Torres-Cueco R, Albornoz-Verdugo M, Guzman-Munoz E. Update on the effects of graded motor imagery and mirror therapy on complex regional pain syndrome type 1: A systematic review. J Back Musculoskelet Rehabil. 2017;30(3):441-449. doi: 10.3233/BMR-150500. PMID 27858687
- [Background] Sawyer EE, McDevitt AW, Louw A, Puentedura EJ, Mintken PE. Use of Pain Neuroscience Education, Tactile Discrimination, and Graded Motor Imagery in an Individual With Frozen Shoulder. J Orthop Sports Phys Ther. 2018 Mar;48(3):174-184. doi: 10.2519/jospt.2018.7716. Epub 2017 Dec 19. PMID 29257926
- [Background] Dilek B, Ayhan C, Yagci G, Yakut Y. Effectiveness of the graded motor imagery to improve hand function in patients with distal radius fracture: A randomized controlled trial. J Hand Ther. 2018 Jan-Mar;31(1):2-9.e1. doi: 10.1016/j.jht.2017.09.004. Epub 2017 Nov 6. PMID 29122370
- [Background] Priganc VW, Stralka SW. Graded motor imagery. J Hand Ther. 2011 Apr-Jun;24(2):164-8; quiz 169. doi: 10.1016/j.jht.2010.11.002. Epub 2011 Feb 9. PMID 21306870
- [Background] Birinci T, Razak Ozdincler A, Altun S, Kural C. A structured exercise programme combined with proprioceptive neuromuscular facilitation stretching or static stretching in posttraumatic stiffness of the elbow: a randomized controlled trial. Clin Rehabil. 2019 Feb;33(2):241-252. doi: 10.1177/0269215518802886. Epub 2018 Oct 10. PMID 30304958
- See also: Graded Motor Imagery — http://www.gradedmotorimagery.com/